CLINICAL TRIAL: NCT00717574
Title: Addition of Nitrous Oxide to a Sevoflurane or Propofol Based Anesthetic and Its Effects on Depth of Anesthesia Indices (N20)
Brief Title: Addition of Nitrous Oxide and Its Effects on Depth of Anesthesia
Acronym: N20
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 13800
Record Dates: First submitted 2008-07-09; First posted 2008-07-17 (Estimated); Results first posted 2017-06-28 (Actual); Last update posted 2017-07-31 (Actual); Status verified 2017-06

CONDITIONS: Deep Sedation; Anesthesia, General
Keywords: depth of sedation; nitrous oxide; general anesthesia; anesthesia indices
MeSH Terms: interventions — Nitrous Oxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sevoflurane group (Active Comparator): Sevoflurane based general anesthesia
  Interventions: Drug: Sevoflurane group
- Propofol group (Active Comparator): Propofol based general anesthesia
  Interventions: Drug: Propofol group

INTERVENTIONS:
Drug: Sevoflurane group — Addition of 60% nitrous oxide for 20 minutes duration, then back to 1:1 oxygen/air mixture.
  Other Names: nitrous oxide
  Arms: Sevoflurane group
Drug: Propofol group — Addition of 60% nitrous oxide for 20 minutes duration, then back to 1:1 oxygen/air mixture.
  Other Names: nitrous oxide
  Arms: Propofol group

SUMMARY:
The study hypothesizes that adding 60% nitrous oxide to a steady state sevoflurance or propofol anesthetic will lead to a decrease in both BIS and Entropy indices during a constant level of surgical stimulus

DETAILED DESCRIPTION:
Nitrous oxide is a widely used general anesthetic pas. It is often used in addition to a second, more potent agent. BIS and Entropy are depth of anesthesia monitors in clinical use. There are conflicting reports about the usefulness of these monitors when nitrous oxide is used as a part of the anesthetic regimen. While some studies demonstrate a decrease in BIS and Entropy, this study aims to investigate the effects of adding nitrous oxide to a sevoflurane or a propofol based anesthetic on BIS and Entropy indices.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18 to 55yrs
* ASA status less than and equal to 2

Exclusion Criteria:

* Surgery on head and neck
* ASA greater than 3
* Contraindication to nitrous oxide
* Pregnant women
* History of dementia and stroke, or other organic brain disorder
* Prisoner
* Ear surgery

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2008-03; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet S Ozcan, M.D., Principal Investigator — Univeristy of Illinois Chicago
Locations (1):
- University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Anderson RE, Jakobsson JG. Entropy of EEG during anaesthetic induction: a comparative study with propofol or nitrous oxide as sole agent. Br J Anaesth. 2004 Feb;92(2):167-70. doi: 10.1093/bja/aeh036. PMID 14722164

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study includes patients aged 18 to 55 years who were classified as ASA physical status ≤2 and scheduled to have surgery under general anesthesia . Only patients for which intraoperative Entropy or BIS monitoring was planned were enrolled by speaking to the attending anesthesiologists working at the OU Presbyterian hospital.
Pre-assignment Details: Patients were randomized into 2 groups that differ in the choice of the agent for the maintenance of general anesthesia: sevoflurane or propofol.
Period: Overall Study
Arm/Group | Sevoflurane Group | Propofol Group
Started | 16 | 16
Completed | 14 | 14
Not Completed | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sevoflurane Group | Propofol Group | Total
Number analyzed (Participants) | 14 | 14 | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 39 (10) | 38 (9.6) | 38.7 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 10 | 18
  Male | 6 | 4 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 3 | 5
  White | 9 | 10 | 19
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 14 | 14 | 28
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 31 (6) | 32 (10) | 31.5 (8)

OUTCOME MEASURES:

1. Primary Outcome: The Effect of Nitrous Oxide on Bispectral Index (BIS) and State Entropy Index (SE)
Description: We planned this study to compare the effect of adding N2O on BIS and SE during an intravenous or an inhalation anesthetic. We hypothesized that neither BIS nor SE would decrease in response to the addition of N2O to a Propofol anesthetic. We also hypothesized that neither BIS nor SE would decrease in participants under Sevoflurane anesthesia if the inspired concentration of Sevoflurane were carefully and continuously adjusted to maintain a constant end-tidal concentration during the addition and discontinuation of N2O.
  BIS (0-100) and SE (0-92) are unitless, ordinal indices of anesthetic depth. Both indices are decreased when the depth of anesthesia is increased.
Time Frame: From baseline to 20 minutes after the addition of 60% nitrous oxide
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sevoflurane Group | Propofol Group
Number analyzed (Participants) | 14 | 14
units on a scale
  Baseline BIS | 36 (7) | 40 (10)
  60% Nitrous Oxide BIS | 32 (7) | 39 (10)
  Baseline SE | 37 (10) | 43 (11)
  60% Nitrous Oxide SE | 31 (11) | 43 (12)

ADVERSE EVENTS:
Time Frame: Patients were monitored for the adverse event from start of the surgery until the patient was discharged from the post anesthesia care unit.
Arm/Group | Sevoflurane Group | Propofol Group
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 0/14 | 0/14

LIMITATIONS AND CAVEATS:
1. We did not measure the blood concentrations of Sevoflurane.
2. Variety of surgical procedures might have lead to different levels of noxious stimuli.
3. Noxious stimuli and administration of opioids may affect EEG-derived indices.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No